CLINICAL TRIAL: NCT06439173
Title: Study of the Hematopoietic Niche and the Role of Inflammation in the Pathophysiology of Cytopenias After CAR-T Cell Therapy: Potential of Therapies Directed to Repair the Bone Marrow Microenvironment
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: PI23/01107; PI2024 03 1552 (Registry Identifier: Ethics Committee for Drug Research of the Salamanca Health Area)
Record Dates: First submitted 2024-04-18; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Lymphoma B Cell; CAR-T Therapy; Cytopenia; Hematopoietic Niche; Inflammation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Cytopenia; Inflammation | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: CAR-T cell therapy — Patients with diffuse large B-cell lymphoma undergoing consecutive commercial CAR-T therapy at the University Hospital of Salamanca

SUMMARY:
Immunotherapy with chimeric antigen receptor T-cells (CAR-T) has revolutionized the treatment of oncohematological diseases and its applications in solid tumors and non-neoplastic diseases are advancing. Cytopenias after CAR-T therapy are the most frequent complication in the medium and long term after treatment, they are a cause of morbimortality, and there are no effective therapies available.

The general objective of the present research project is to analyze, in a series of 40 patients with diffuse large B-cell lymphoma undergoing consecutive commercial CAR-T therapy at the University Hospital of Salamanca, the characteristics of the hematopoietic niche and the systemic and bone marrow inflammatory status in patients with prolonged cytopenias after CAR-T cell therapy with respect to those without cytopenias and with respect to the pre-treatment situation (performing quantitative and functional analysis of the stroma by immunohistochemistry, flow cytometry and genomic studies, in addition to functional hematopoietic assays-clonogenic assays, long-term cultures-), and to evaluate both in vitro (by co-culturing with macrophages activated by CAR-T/tumor cell interaction and assessing cytokines) and in vivo (in an animal model of lymphoma and CRS) the therapeutic potential of therapies aimed at repairing the hematopoietic bone marrow microenvironment, such as the use of allogeneic mesenchymal cells (MSC) from healthy donors and MSC-derived extracellular vesicles (MSC-EV) studying their effects on inflammatory mediators, hematopoiesis and the cytotoxic effect of CAR-T.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diffuse large B-cell lymphoma undergoing consecutive commercial CAR-T therapy
* Over 18 years old
* Sign the informed consent

Exclusion Criteria:

* Under 18 years old
* Do not sign the informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with diffuse large B-cell lymphoma undergoing consecutive commercial CAR-T therapy at the University Hospital of Salamanca
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterizing hematopoietic niche post CAR-T Therapy | 36 months
  To analyze the characteristics of the hematopoietic niche in patients experiencing prolonged cytopenias post CAR-T cell therapy compared to those without cytopenias and their pre-treatment status.
Characterizing systemic inflammation post CAR-T Therapy | 36 months
  To analyze the characteristics of systemic inflammatory status in patients experiencing prolonged cytopenias post CAR-T cell therapy compared to those without cytopenias and their pre-treatment status.
Characterizing medullary inflammation post CAR-T Therapy | 36 months
  To analyze the characteristics of medullary inflammatory status in patients experiencing prolonged cytopenias post CAR-T cell therapy compared to those without cytopenias and their pre-treatment status.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Asistencial Universitario de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided